CLINICAL TRIAL: NCT00906867
Title: Pulmonary Function Test, Bronchial Hyperresponsiveness and Quality of Life in Patients With Vocal Cord Dysfunction (VCD)
Acronym: VCD
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Johannes Schulze MD, Cosultant Pediatric Allergy and Pulmonolgy, Johann Wolfgang Goethe University Hospital
Other Study IDs: KGU-62/09
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Dyspnea
Keywords: Vocal cord dysfunction; Laryngoscopy; Methacholine challenge; Pulmonary function testing
MeSH Terms: conditions — Dyspnea; Vocal Cord Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum, total IgE
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vocal cord dysfunction: Patients with suspicion of VCD
  Interventions: Other: Methacholine challenge testing; Procedure: Rhino-laryngoscopy

INTERVENTIONS:
Other: Methacholine challenge testing — Nebulized methacholine administered at the following doses: 0,1 mg/0,4 mg/0,8 mg/1,6 mg
  Other Names: Aerosol Provocation System (Cardinal Health GmbH)
Procedure: Rhino-laryngoscopy — Topical anesthesia (Xylocain Pump spray) followed by transnasal fiberoptic laryngoscopy with a flexible fiberoptic laryngoscope.
  Other Names: ENF-V2 laryngoscope Olympus

SUMMARY:
Vocal cord dysfunction is a rare clinical picture. It is labeled as a sudden and threatening dyspnea. Patients with VCD may also present cough, hoarseness, wheezing, and chest tightness, but an inspiratory stridor is the most common symptom. For this reason, such patients are often misdiagnosed with refractory asthma, because of poor response to steroids and bronchodilators. Diagnosis is suspected on clinical grounds and is confirmed with laryngoscopy. The therapy consists of education, speech therapy and if necessary psychotherapy. The purpose of the investigators' study is to characterize children, adolescents, and young adults with VCD, and the evaluation of predictors as atopy, bronchial hyperresponsiveness, and psychiatric features.

DETAILED DESCRIPTION:
VCD appears to be significantly more common among females. The episode of dyspnea underlies the paradoxical, intermittent adduction of the vocal cords during inspiration. Methacholine challenge testing combined with laryngoscopy is useful in differentiating vocal cord dysfunction from asthma during the asymptomatic period.

In one visit patients will be characterized with a questionnaire based on the ISAAC questionnaire. Furthermore, FeNO, eCO, skin prick testing and total serum IgE will be examined. The psychiatric condition of patients will be determined by CBCL/6-18 and YSR/11-18 behavior questionnaires. After initial fiberoptic laryngoscopy and pulmonary function testing, bronchoprovocation is performed using nebulized methacholine at increasing doses, until a 20% decline in the forced expiratory volume in 1 second is achieved (PD20FEV1). Each methacholine testing will be followed by a second laryngoscopy and pulmonary function testing. The visualization of paradoxical vocal cord motion during inspiration will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 7 to 30 Years
* Documented VCD or strong suspicion of VCD
* Pulmonary function test: FEV1 (% pred.) ≥ 70%

Exclusion Criteria:

* Age < 7 and > 30 Years
* Pulmonary function test: FEV1 (% pred.) < 70%
* Others chronic diseases or infections (e.g., HIV, tuberculosis, malignancy)
* Pregnancy
* Documented alcohol, substance, and/or drug abuse
* Incapability to perform all study procedure
* Current participation in another clinical trial

Ages: 7 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Outpatients of departement of Pediatric Pulmonology and Allergology.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Characterization of vocal cord dysfunction, and evaluation of predictors as atopy, bronchial hyperresponsiveness, and psychiatric behavior. | one day

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, Prof, Principal Investigator — Goethe University, Frankfurt, Germany
Locations (1):
- Goethe University Hospital, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Perkins PJ, Morris MJ. Vocal cord dysfunction induced by methacholine challenge testing. Chest. 2002 Dec;122(6):1988-93. doi: 10.1378/chest.122.6.1988. PMID 12475837
- [Background] Guss J, Mirza N. Methacholine challenge testing in the diagnosis of paradoxical vocal fold motion. Laryngoscope. 2006 Sep;116(9):1558-61. doi: 10.1097/01.mlg.0000228007.74561.33. PMID 16954978
- [Background] Husein OF, Husein TN, Gardner R, Chiang T, Larson DG, Obert K, Thompson J, Trudeau MD, Dell DM, Forrest LA. Formal psychological testing in patients with paradoxical vocal fold dysfunction. Laryngoscope. 2008 Apr;118(4):740-7. doi: 10.1097/MLG.0b013e31815ed13a. PMID 18182970
- [Background] Sandage MJ, Zelazny SK. Paradoxical vocal fold motion in children and adolescents. Lang Speech Hear Serv Sch. 2004 Oct;35(4):353-62. doi: 10.1044/0161-1461(2004/034). PMID 15609638
- [Background] Loughlin CJ, Koufman JA. Paroxysmal laryngospasm secondary to gastroesophageal reflux. Laryngoscope. 1996 Dec;106(12 Pt 1):1502-5. doi: 10.1097/00005537-199612000-00011. PMID 8948611
- [Background] Newman KB, Mason UG 3rd, Schmaling KB. Clinical features of vocal cord dysfunction. Am J Respir Crit Care Med. 1995 Oct;152(4 Pt 1):1382-6. doi: 10.1164/ajrccm.152.4.7551399.
- [Background] Mikita CP, Mikita JA. Allergic bronchopulmonary aspergillosis. Allergy Asthma Proc. 2006 Jan-Feb;27(1):82-4. PMID 16598999
- [Background] Crapo RO, Casaburi R, Coates AL, Enright PL, Hankinson JL, Irvin CG, MacIntyre NR, McKay RT, Wanger JS, Anderson SD, Cockcroft DW, Fish JE, Sterk PJ. Guidelines for methacholine and exercise challenge testing-1999. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. Am J Respir Crit Care Med. 2000 Jan;161(1):309-29. doi: 10.1164/ajrccm.161.1.ats11-99. No abstract available. PMID 10619836
- [Background] Asher MI, Keil U, Anderson HR, Beasley R, Crane J, Martinez F, Mitchell EA, Pearce N, Sibbald B, Stewart AW, et al. International Study of Asthma and Allergies in Childhood (ISAAC): rationale and methods. Eur Respir J. 1995 Mar;8(3):483-91. doi: 10.1183/09031936.95.08030483. PMID 7789502